CLINICAL TRIAL: NCT01626768
Title: Medtronic Market-Released DF4 Lead Imaging
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: DF4-Imaging-2012
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Tachycardia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled patients

SUMMARY:
The Medtronic Market-Released DF4 Lead Imaging Study is a prospective, non-randomized study, multi-center clinical investigation.

The purpose of this clinical investigation is to collect high quality medical images of the Medtronic Market-Released DF4 lead in the shoulder and heart. Images collected during the study will allow for lead design and testing processes better tailored to the implanted environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age.
* Patients able and willing to attend imaging session.
* Patients able and willing to give informed consent.
* Patients with an implanted device/lead(s) for a minimum of 3 months.

Exclusion Criteria:

* Subjects who require a legally authorized representative to obtain consent.
* Subjects with exclusion criteria required by local law (e.g. age, breastfeeding
* Pregnant women, or women of child bearing potential and who are not on a reliable form of birth control.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
In vivo lead shape | Six Months

CONTACTS AND LOCATIONS:
Locations (2):
- Riyadh, Saudi Arabia
- London, United Kingdom